CLINICAL TRIAL: NCT04147910
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-KW-6356 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-KW-6356
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6356-009
Record Dates: First submitted 2019-10-09; First posted 2019-11-01 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Healthy Male Subjects
Keywords: Healthy Male Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KW-6356 (Experimental): Single oral dose of carbon-14-KW-6356.
  Interventions: Drug: KW-6356

INTERVENTIONS:
Drug: KW-6356 — Single oral dose of KW-6356

SUMMARY:
This is an open-label, single-dose study in healthy male subjects to investigate the absorption, metabolism, and excretion (AME) of KW-6356.

DETAILED DESCRIPTION:
Subjects will be screened to assess their eligibility to enter the study within approximately 4 weeks prior to dose administration. Subjects will be confined to the Clinical Research Unit (CRU) for their entire participation in this study. Eight subjects will be enrolled to allow 6 subjects to complete the study. Each subject will report to the CRU and be confined from Day -1 (the day before dosing) through at least Day 8 (168 hours postdose). A single dose of study drug will be administered on Day 1 (0 hour). On Day 8, subjects can be asked to remain as a resident within the CRU for an additional period to allow for ongoing 24-hour urine, fecal, and blood sample collections. These collections can continue up to a maximum of 336 hours postdose (Day 15). Subjects can be discharged prior to Day 15 if the following individual subject discharge criteria have been satisfied: ≥ 90% of the 14C dose recovered in combined urine and feces, and ≤ 1% of the total radioactive dose is recovered in combined excreta (urine and feces) in 3 consecutive 24-hour periods in which a fecal sample is provided.

ELIGIBILITY:
Inclusion Criteria:

1. Males, of any race, between 18 and 65 years of age, inclusive.
2. Body mass index between 18.0 and 30.0 kg/m2, inclusive.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital sign measurements, and clinical laboratory evaluations.
4. Able to sign an ICF and willing to abide by the study restrictions.
5. Will agree to use contraception.
6. History of at least 1 bowel movement per day.

Exclusion Criteria:

1. Any clinically significant illness as determined by the Principal Investigator.
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance.
3. Have received any investigational drug within 30 days or 5.5 half-lives, whichever is longer, prior to study dosing.
4. History of drug or alcohol abuse or dependence within 2 years prior to signing of ICF.
5. Hospital admission, surgery, within 3 months before investigational product administration.
6. Positive hepatitis B surface antigen or hepatitis C RNA, or positive for acquired human immunodeficiency virus.
7. Positive urine drug screen for drugs of abuse.
8. History of requiring treatment for urinary retention within 3 months before investigational product administration.
9. History of seizures.
10. Subjects with history of, or active suicidal ideation, or suicide attempt.
11. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed). Subjects with cholecystectomy will not be allowed.
12. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including inducers/inhibitors of CYP3A4 and St. John's wort, within 30 days prior to Day 1.
13. Use or intend to use any prescription medications/products within 30 days or 5.5 half-lives (if known), whichever is longer, prior to Check-in.
14. Use or intend to use slow-release medications/products considered to still be active within 30 days or 5.5 half-lives (if known), whichever is longer, prior to Check-in.
15. Use of any nonprescription medications (for 14 days prior to Check-in).
16. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in, or positive cotinine.
17. Receipt of blood products within 2 months prior to Check-in.
18. Donation of blood (> 200 mL) from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
19. Poor peripheral venous access.
20. Have previously completed or withdrawn from this study or any other study investigating KW-6356, and have previously received the investigational product.
21. Subjects with exposure to significant diagnostic or therapeutic radiation (eg, serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in.
22. Subjects who have participated in a radiolabeled drug study where exposures are known to the Investigator within the previous 4 months prior to admission to the clinic for this study or participated in a radiolabeled drug study where exposures are not known to the Investigator within the previous 6 months prior to admission to the clinic for this study.
23. Subjects who, in the opinion of the Investigator, should not participate in this study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Maximum observed concentration (KW-6356 in plasma and total radioactivity in plasma and blood).
tmax | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Time of maximum observed concentration (KW-6356 in plasma and total radioactivity in plasma and blood).
AUC0-t | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Area under the drug concentration-time curve from time zero to the last quantifiable concentration (KW-6356 in plasma and total radioactivity in plasma and blood).
%AUCextra | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Percentage of estimated part for the calculation of AUC0-∞ (KW-6356 in plasma and total radioactivity in plasma and blood).
t1/2 | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Elimination half-life (KW-6356 in plasma and total radioactivity in plasma and blood).
kel | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Elimination rate constant (KW-6356 in plasma and total radioactivity in plasma and blood).
Vz/F | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Apparent volume of distribution during terminal phase (KW-6356 in plasma).
CL/F | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Apparent oral clearance (KW-6356 in plasma).
MRT | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Mean residence time (KW-6356 in plasma).
Whole blood/plasma concentration ratio (total radioactivity in blood and plasma). | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
Aeurine | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Cumulative amount excreted in urine (total radioactivity in urine).
feurine | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Fraction of the dose administered excreted in urine (total radioactivity in urine).
Aefeces | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Cumulative amount excreted in feces (total radioactivity in feces).
fefeces | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Fraction of the dose administered excreted in feces (total radioactivity in feces).
Aetotal | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Total amount excreted (total radioactivity in urine and feces).
fetotal | Pre-dose up to 168 hours post dose, up to 336 hours post dose.
  Fraction of the dose administered excreted in urine and feces (total radioactivity in urine and feces).
Metabolic profiling and identification (plasma, urine, and feces). | Pre-dose up to 168 hours post dose, up to 336 hours post dose.

SECONDARY OUTCOMES:
Adverse Events | From screening through study completion, an average of 6 weeks.
  Number of subjects experiencing an adverse event related to treatment.
Severe adverse events. | From screening through study completion, an average of 6 weeks.
  Number of subjects experiencing a severe adverse event related to treatment.
Serum chemistry, hematology, and urinalysis. | From screening through study completion, an average of 6 weeks.
  Number of subjects with abnormal laboratory values that are related to treatment.
Vital signs | From screening through study completion, an average of 6 weeks.
  Number of subjects with abnormal vital signs that are related to treatment.
12-lead ECG. | From screening through study completion, an average of 6 weeks.
  Number of subjects with abnormal ECG that are related to treatment.
Physical examination. | From screening through study completion, an average of 6 weeks.
  Number of subjects with abnormal physical exam findings that are related to treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No